CLINICAL TRIAL: NCT01927393
Title: Integration of Palliative Care Planning in Pancreatic and Ovarian Cancers
Brief Title: Palliative Care in Improving Quality of Life and Symptoms in Patients With Stage III-IV Pancreatic or Ovarian Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not funded
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13270; NCI-2013-01629 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13270 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2013-08-20; First posted 2013-08-22 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IIIA Ovarian Epithelial Cancer; Stage IIIA Ovarian Germ Cell Tumor; Stage IIIB Ovarian Epithelial Cancer; Stage IIIB Ovarian Germ Cell Tumor; Stage IIIC Ovarian Epithelial Cancer; Stage IIIC Ovarian Germ Cell Tumor; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Pancreatic Neoplasms | interventions — Palliative Care; Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (PCPI) (Experimental): Patients undergo a comprehensive physical, psychological, social, and spiritual palliative care assessment. Patients also receive a workbook that covers physical and psychological well-being and social and spiritual well-being, delivered over 2 educational sessions.
  Interventions: Other: palliative care; Behavioral: educational intervention; Procedure: quality-of-life assessment; Other: questionnaire administration
- Arm II (standard care plus attention control) (Active Comparator): Patients receive standard care plus attention comprising two telephone contacts.
  Interventions: Procedure: quality-of-life assessment; Other: questionnaire administration; Behavioral: telephone-based intervention

INTERVENTIONS:
Other: palliative care — Receive PCPI
  Arms: Arm I (PCPI)
Behavioral: educational intervention — Receive education sessions
  Other Names: intervention, educational
  Arms: Arm I (PCPI)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies
Behavioral: telephone-based intervention — Receive telephone contacts
  Arms: Arm II (standard care plus attention control)

SUMMARY:
This randomized clinical trial studies palliative care in improving quality of life and symptoms in patients with stage III-IV pancreatic or ovarian cancer. Palliative therapy may help patients with advanced pancreatic or ovarian cancer live more comfortably.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the effects of a concurrent palliative care planning intervention (PCPI) on overall quality of life (QOL) and symptom burden.

II. Test the effects of a concurrent PCPI on anxiety and depression. III. Test the effects of a concurrent PCPI on overall survival. IV. Test the effects of a concurrent PCPI on health care resource use.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo a comprehensive physical, psychological, social, and spiritual palliative care assessment. Patients also receive a workbook that covers physical and psychological well-being and social and spiritual well-being, delivered over 2 educational sessions.

ARM II: Patients receive standard care plus attention comprising two telephone contacts.

After completion of study, patients are followed up at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pancreatic or ovarian cancer
* Confirmed stage III or IV disease
* Patients who are within one year from initial diagnosis
* Able to read or understand English-this is included because most of the patient-reported outcome measures are not validated in linguistically diverse populations; the intent is to adapt and test the intervention in a future study with linguistically diverse populations
* Ability to read and/or understand the study protocol requirements, and provide written informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Overall QOL, assessed by the Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) or the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) | Up to 6 months
  The analysis will be a 2x2x3 repeated measures analysis of covariance (ANCOVA) statistical design.
Symptom burden using the FACT-Trial Outcome Index (TOI) | Up to 6 months
  Compared between groups and by diagnoses using two-way contingency table analysis, two way analysis of variance (ANOVA) according to level of measurement.

SECONDARY OUTCOMES:
Reduction in anxiety | Up to 6 months
  Compared demographically by group according to completeness of the intervention using t-tests or one-way ANOVAs according to the level of measurement of the variables. Tested using a 2x2 contingency table analysis and the McNemar test statistic.
Reduction in depression | Up to 6 months
  Compared demographically by group according to completeness of the intervention using t-tests or one-way ANOVAs according to the level of measurement of the variables. Tested using a 2x2 contingency table analysis and the McNemar test statistic.
Overall survival | At 6 months
  Compared demographically by group according to completeness of the intervention using t-tests or one-way ANOVAs according to the level of measurement of the variables.
Health care resource use including presence of advanced care planning, chemotherapy in the last 14 days of life, and length of time between hospice referral and death | Up to 6 months
  Two way (2x2) ANOVAs will be conducted to test the differences between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States